CLINICAL TRIAL: NCT06623669
Title: A Mobile Intervention to Reduce Pain and Improve Health-III
Acronym: MORPH-III
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Wake Forest University Health Sciences (Other); Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Fanning, Assistant Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00025649; R01AG082777 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Osteoarthritis; Obesity and Overweight; Inactivity
Keywords: Digital health; Randomized Trial; Physical Activity; Weight Loss; Aging
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Obesity; Overweight; Sedentary Behavior; Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MORPH (Experimental): MORPH participants will attend one weekly group-mediated session alongside a group of their peers plus individual coaching calls. Participants will aim to increase daily steps by moving often throughout the day, using an activity monitor and mHealth app to view feedback and set goals. Participants will also aim to weight via healthy eating while reducing daily calories by ~400kcal/day below weight maintenance needs to achieve approximately 6% weight loss in 6 months and 10% over 18 months.
  Interventions: Behavioral: MORPH
- Measurement Only (Active Comparator): Measurement-only participants will receive an activity monitor and wireless weight scale to account for the effect of these self-monitoring technologies and activity behavior.
  Interventions: Behavioral: Measurement Only

INTERVENTIONS:
Behavioral: MORPH — A remote behavioral intervention combining coaching and digital health tools to improve diet and activity behaviors.
  Arms: MORPH
Behavioral: Measurement Only — This intervention entails receipt of a body weight scale and wearable activity monitor.
  Arms: Measurement Only

SUMMARY:
The experience of chronic pain powerfully and negatively affects quality of life and functional independence in aging. Unfortunately, while as many as three in four older adults experience chronic pain, few have access to effective non-pharmacological pain management strategies. Participating in regular physical activity, avoiding sustained sitting, and maintaining a healthy weight are important and interrelated lifestyle inputs to chronic pain, and socially rich behavioral interventions informed by contemporary theories of behavior change appear important for engaging in activity and healthy eating in the long term. Our group has demonstrated in a series of Stage I trials that a group-mediated behavioral intervention combining dietary behavior change and a physical activity program focused on moving often throughout the day contributes to meaningful weight loss, and lasting weight maintenance, with pilot data suggesting this may contribute to improved pain, physical function, and health-related quality of life among older adults with chronic pain. As these were NIH Stage I trials, there are several important gaps to be addressed in the present trial: (1) both studies of chronic pain recruited small samples and were 12 weeks in duration, limiting our ability to establish efficacy and the durability of changes to activity, HRQOL, and pain outcomes; (2) participants included anyone with chronic pain, regardless of pain type, a likely contributor to heterogeneous pain intensity and interference findings; and (3) the investigators have yet to examine behavioral maintenance.

The overarching goal of the proposed Stage II "mobile intervention to reduce pain and improve health-III (MORPH-III)" is to establish the efficacy of the intervention for enhancing physical activity via steps (primary), and for reducing pain interference and body weight while enhancing physical function (secondary) among older adults with chronic knee or hip osteoarthritic (OA) pain. The investigators will recruit 200 older adults with knee or hip osteoarthritic pain to engage in a 6-month remotely delivered intervention comprising weekly group or individual intervention meetings plus brief individual goal-setting coaching calls. This will be followed by a 12-month no-contact maintenance period, where participants will attempt to sustain behavioral goals on their own.

The Specific Aims are:

Specific Aim 1: To examine the impact of MORPH on ActivPAL-assessed daily steps relative to an enhanced usual care control. Hypotheses: MORPH will significantly increase steps relative to control at month 6.

Specific Aim 2: To examine the impact of MORPH on pain interference, change in body weight, and physical function relative to the enhanced usual care control. Hypotheses: MORPH will result in significant reductions in pain interference and body weight and improvement in physical function relative to control at month 6.

Exploratory Aims: Aim 1: To investigate the impact of the MORPH intervention on steps, weight change, pain interference, and physical function at month 18. Aim 2: If the MORPH intervention results in reduced pain interference at 6 and/or 18 months, the investigators will examine the extent to which 6-month change in steps, weight, pain self-efficacy, and catastrophizing mediate change in interference at 6 and/or 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65+ years
* Body mass index of 30-45 kg/m2 or >45 kg/m2 with physician's approval
* No loss or gain of more than 5% body mass in previous 6 months
* Presence of knee or hip osteoarthritis as ascertained via the Roux questionnaire
* Independently living
* Low active (i.e., not participating in regular resistance training and/or >20 mins/day of aerobic exercise on more than 2 days/week in past 3 months as ascertained via a modified CHAMPS questionnaire)
* Have no contraindication for safe and optimal participation in exercise based on EASY screening
* Not currently using a weight loss medication
* Approved for participation by medical director
* Willing to provide informed consent and agree to all study procedures and assessments.

Exclusion Criteria:

* Reside in skilled nursing facility, rehab or assisted living environment
* History of pharmacologic treatment for a psychiatric disorder other than depression/anxiety within past year
* Current untreated and/or unstable clinical depression or anxiety (Patient Health Questionnaire (PHQ-9) >15)
* Hospitalization for psychiatric event within past year prior to screening
* History of mild cognitive impairment or dementia
* Cognitive impairment (<32) on Modified Telephone Interview for Cognitive Status survey (TICS-M)
* Hearing or visual impairment that would preclude use of the videoconferencing software
* Severe arthritis or other musculoskeletal disorder that is a contraindication for safe walking
* Presently undergoing treatment for orthopedic fracture
* Currently using a weight loss medication
* Contraindication based on EASY screening without physician approval.
* Joint replacement or other orthopedic surgery in past 6 months
* Joint replacement or other orthopedic surgery planned in next 18 months
* Have a diagnosis of uncontrolled hypertension; current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease other than asthma or COPD, any disease requiring oxygen use, neurological or hematological disease; cancer requiring current treatment, except non-melanoma skin cancers; kidney failure requiring dialysis; have a Katz ADL disability; or engage in heavy alcohol use >14 drinks/week.
* Current participation in other research study with a prospective intervention
* Unable/unwilling to commit to study protocol, including random assignment and use of technology tools
* Unable/unwilling to attend three virtual testing appointments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Daily steps | Baseline, after 6 months of intervention, after 18 months of intervention
  Daily steps measured over one week via the ActivPAL accelerometer

SECONDARY OUTCOMES:
Pain Interference | Baseline, after 6 months of intervention, after 18 months of intervention
  Measured via questionnaire: the Patient-Reported Outcomes Measurement Information System (PROMIS) 8-item pain interference scale, which produces a t-score such that the population mean is a 50 with a standard deviation of 10; higher scores indicate higher interference.
Body weight | From the start of the intervention through month 18.
  Measured via the BodyTrace wireless body weight scale
30-second chair stand | Baseline, after 6 months of intervention, after 18 months of intervention
  Measured via in-home chair stand task.
Gait speed | Baseline, after 6 months of intervention, after 18 months of intervention
  Measured via in-home test: 4-meter habitual gait speed

OTHER OUTCOMES:
Physical activity behavior | Collected over one week at baseline, after 6 months of intervention, after 18 months of intervention
  Directly measured using the ActivPAL 4 accelerometer
Adverse Events | Baseline, after 6 months of intervention, after 18 months of intervention
  Assessed via assessor query and spontaneous report
Participant Feedback | After 6 months of intervention
  Assessed via semi-structured interview
Medication usage | Baseline, after 6 months of intervention, after 18 months of intervention
  Assessed via assessor query
Sleep behavior | Nightly over the 18-month intervention
  Assessed via wearable activity monitor
Pain intensity | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the 3-item Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale, which produces a t-score such that the population mean is a 50 with a standard deviation of 10; higher scores indicate higher interference.
Perceived physical function | Baseline, after 6 months of intervention, after 18 months of intervention.
  Self-Reported via the Pepper Assessment Tool for Disability. The scale produces a total score and subscales capturing basic activities of daily living, mobility, and instrumental activities of daily living. Scores range from 1-6 with lower scores representing less disability.
Pain Catastrophizing | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Pain Catastrophizing Scale. The scale produces a total score (range 0 - 52) and subscales including rumination (range 0 - 16), magnification (range 0 - 12), and helplessness (range 0 - 24). Higher scores represent greater catastrophizing.
Self-determinative needs | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Basic Psychological Need Satisfaction and Frustration Scales. Produces six subscale scores: autonomy satisfaction and frustration, relatedness satisfaction and frustration, and competence satisfaction and frustration. Scores for each subscale range from 4 - 20 such that higher scores represent greater satisfaction or frustration.
Affect | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Positive and Negative Affect Schedule. The scale produces a positive affect score and a negative affect score, which each range from 10 - 50 whereby higher scores indicate greater positive or negative affect.
Stress | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the 10-item perceived stress scale. Scores range from 0 - 40 with higher scores indicating greater stress.
Exercise Self-Efficacy | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Exercise Self-Efficacy Scale as well as by a modified version of the scale to capture accumulated physical activities. Final scores range from 0 - 100 with higher scores reflecting greater self-efficacy.
Outcome Expectencies related to Eating Behavior | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Outcome Expectations for Nutrition Scale. The scale produces subscales for physical, social, and self-evaluative outcome expectancies with scores range from 5-25. Higher scores reflect more positive expectations in each domain.
Outcome Expectencies related to Activity Behavior | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Outcome Expectations for Exercise Scale, modified to capture all daily physical activities. The scale produces subscales for physical, social, and self-evaluative outcome expectancies with scores range from 5-25. Higher scores reflect more positive expectations in each domain.
Self-regulation | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Self-Regulation Strategy Usage for Nutrition and Activity. The scales produce scores for nutrition and activity behaviors, which each range from 10-50 such that higher scores reflect greater self-regulation strategy usage.
Barriers | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Perceived Barriers for Physical Activity and Eating. The scales produce scores for eating and activity behaviors, with each ranging from 1 - 5 such that higher scores indicate more barriers.
Health-related quality of life | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the 36-item Short Form Health Survey (SF36). Scores are generated for 8 subdomains (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health). Scores for each subscale range from 0 - 100; higher scores are better.
Perceived Sleep | Baseline, after 6 months of intervention, after 18 months of intervention
  Self-reported using the Pittsburgh Sleep Quality Index. The scale yields a total score of 0 - 21 such that 0 represents no sleep difficulty and 21 represents severe difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fanning, PhD, Principal Investigator — Wake Forest University; Amber Brooks, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available via the Wake Forest Pepper Center Study Registry for the outcome measures described in the Outcome Measures section.
Supporting Information: Study Protocol
Time Frame: The research community will have access to the data at the end of the performance period or the time of an associated publication (whichever is earlier). Data will be made available within the Pepper Study Registry in perpetuity.
Access Criteria: Data will be available for investigators providing an Institutional Review Board (IRB)/Ethics approval or certification of exemption from IRB/Ethics review and agreeing to the terms and conditions of a data use agreement. To request access to the data, researchers will use the standard processes for the repository where the data are deposited. This involves user registration, which includes a requirement to review and agree to Terms of Service, ensuring that study data will be used for scholarly scientific research, that data will not be shared with others outside of those listed on a given project proposal, that the data will be presented in aggregate, that researchers will not attempt to present individual data or attempt to identify individuals, and that any potential identification is immediately disclosed.